CLINICAL TRIAL: NCT00940628
Title: Open-label Comparative Randomized Study of the Efficacy and Safety of Orlistat (Xenical) in Complex Therapy of Obesity and Metabolic Disorders in Adolescents
Brief Title: A Study of Xenical (Orlistat) in Overweight and Obese Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: ML19569
Record Dates: First submitted 2009-06-16; First posted 2009-07-16 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet; Exercise; Orlistat

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Diet and Exercise; Drug: orlistat [Xenical]
- 2 (Other)
  Interventions: Behavioral: Diet and Exercise

INTERVENTIONS:
Behavioral: Diet and Exercise — mildly hypocaloric diet and physical exercise
Drug: orlistat [Xenical] — 120mg po tid
  Arms: 1

SUMMARY:
This 2 arm study will assess the effect of Xenical on body mass index (BMI)in obese or overweight adolescents. Patients will be randomised into one of 2 groups; both groups will undergo a regimen of mildly hypocaloric diet and physical exercise, but one group will also receive Xenical 120mg po tid. The anticipated time on study treatment is 1 year, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adolescent patients, 12-14 years of age
* overweight or obese

Exclusion Criteria:

* age <12 or >14 years
* BMI in normal range

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in BMI | At each clinic visit, every 4 weeks

SECONDARY OUTCOMES:
Adverse events, laboratory parameters | At each clinic visit, every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Russia (11):
  - Kazan'
  - Khabarovsk
  - Krasnodar
  - Krasnoyarsk
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Samara
  - Tyumen
  - Yaroslavl
  - Yekaterinburg